CLINICAL TRIAL: NCT04852224
Title: Strength, Aging, and Memory in Prostate Cancer: A Prospective Study of the Effects of Androgen Deprivation on Neurocognition and Frailty
Brief Title: Strength, Aging, and Memory in Prostate Cancer
Acronym: STAMP
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: American College of Sports Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 0261-21-FB
Record Dates: First submitted 2021-04-15; First posted 2021-04-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Prostate Neoplasm; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Androgen Deprivation Therapy (ADT+): Men diagnosed with prostate cancer and scheduled to receive greater than or equal to 6-months of treatment with androgen deprivation therapy
- Prostate Cancer Surveillance (ADT-): Men diagnosed with prostate cancer under active surveillance (i.e., not receiving active treatment for prostate cancer)
- Non-cancer Control (PCa-): Age-matched men without a history of cancer

SUMMARY:
The objective of this study is to compare changes in neurocognitive function across a 12-month period between three groups: (1) men treated with androgen deprivation therapy (ADT) for prostate cancer (PCa); (2) men under active surveillance for PCa; and (3) men without a history of cancer.

DETAILED DESCRIPTION:
Aim 1: This study will examine differences in neurocognitive function (cognitive performance, brain structural integrity) from baseline (within 30 days of ADT initiation or 90 days of diagnosis) to 6- and 12-month follow-up.

Aim 2: Examine group differences in components of frailty (e.g., lean mass, muscle strength, physical function, fatigue, physical activity) from baseline to 6- and 12-month follow-up.

Men will be recruited for this study if they are (1) recently diagnosed with PCa and scheduled to receive 6-months or more of ADT (ADT+ group, n=20), (2) recently diagnosed with PCa and under active surveillance (ADT- group, n=20), or (3) healthy men without a history of cancer (PCa- group, n=20). Eligible men (N=60) will be scheduled for two or three testing appointments at each testing timepoint. To assess Aim 1, participants will complete measures at baseline (M0), 6-month follow-up (M6), and 12-month follow-up (M12). Aim 1 measures include: neurocognitive tasks, functional magnetic resonance imaging (optional; n=10 ADT+ and n=10 ADT- only), and questionnaires. To assess Aim 2, outcomes indicated as components of frailty syndrome will be measured, including: dual-energy X-ray absorptiometry (e.g., appendicular lean mass), upper and lower body dynamometry, physical function and functional capacity, questionnaires (i.e., fatigue surveys), and physical activity monitoring (i.e., accelerometry). Findings from this study will build upon the scientific framework for the potential frailty pathway of cancer-associated cognitive decline in PCa patients in order to develop future evidence-based interventions to manage cognitive impairment in men diagnosed with PCa.

ELIGIBILITY:
Inclusion Criteria:

* Telephone Interview of Cognitive Status (TICS-M) performance above impaired range (≥21)

Group-specific criteria:

* First time, primary diagnosis of prostate cancer (ADT+ and ADT-)
* Diagnosed within past 30 days (ADT-)
* Scheduled to receive ≥ 6-months androgen deprivation therapy and have not received >30 days of androgen deprivation therapy (ADT+)
* Men without a history of cancer who are within one year of age of ADT+ participants (PCa-)

Exclusion Criteria:

* Second cancer diagnosis (excluding non-invasive skin cancers)
* History of stroke, transient ischemic attack, neurological disorder, or brain surgery involving tissue removal
* Unable to walk without assistance
* Unwilling to complete study requirements
* Body weight greater than 300 pounds (DXA requirement)
* Moderate-intensity physical activity ≥ 150 minutes per week
* Upper and lower body strength training ≥ 2 days per week
* Unable to read in English

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men aged 19 years and older diagnosed with prostate cancer either under active surveillance or scheduled to receive/within 30 days of receiving androgen deprivation therapy; and age-matched men without a history of cancer.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Change in inhibitory control | Baseline (M0), 6-month follow-up (M6), 12-month follow-up (M12)
  Change in interference score on Stroop task, with negative values indicating lower inhibitory control. The Stroop task interference score is a continuous variable with no minimum or maximum value.
Change in cognitive flexibility | Baseline (M0), 6-month follow-up (M6), 12-month follow-up (M12)
  Change in reaction time on Task-switch task, with higher values indicating lower cognitive flexibility. The Task-switch reaction time is a continuous variable with no minimum or maximum value.
Change in executive function | Baseline (M0), 6-month follow-up (M6), 12-month follow-up (M12)
  Change in completion time on Trails B task, with higher values indicating lower executive function. Trails B completion time is a continuous variable with no minimum or maximum value.
Change in spatial working memory reaction time | Baseline (M0), 6-month follow-up (M6), 12-month follow-up (M12)
  Change in reaction time on spatial working memory task, with faster reaction times indicating better spatial working memory.
Change in short term memory | Baseline (M0), 6-month follow-up (M6), 12-month follow-up (M12)
  Change in accuracy on N-Back task, with higher accuracy indicating better short-term memory.
Change in processing speed | Baseline (M0), 6-month follow-up (M6), 12-month follow-up (M12)
  Change in accuracy on Attentional Blink task, with higher accuracy indicating faster processing speed.
Change in verbal memory | Baseline (M0), 6-month follow-up (M6), 12-month follow-up (M12)
  Change in number recalled on Hopkins Verbal Learning Task, with greater number of items recalled indicating better verbal memory.
Change in visuospatial function | Baseline (M0), 6-month follow-up (M6), 12-month follow-up (M12)
  Change in accuracy on Benton Judgement of Line Orientation task, with higher accuracy indicating better visuospatial function.
Change in white matter integrity | Baseline (M0), 6-month follow-up (M6)
  Change in fractional anisotropy as measured by diffusion MRI.
Change in brain volume | Baseline (M0), 6-month follow-up (M6)
  Change in mean cortical thickness of brain regions of interest as measured by an anatomical MRI brain scan.
Change in resting state functional connectivity | Baseline (M0), 6-month follow-up (M6)
  Change in within-network pairwise correlation estimates as measured using a multiband echo planar imaging (mb-EPI) functional MRI sequence.
Change in self-reported cognitive function | Baseline (M0), 6-month follow-up (M6), 12-month follow-up (M12)
  The perceived cognitive impairments subscale of the Functional Assessment in Cancer Therapy - Cognition (FACT-Cog) will be sued to measure self-reported cognition. Scores range from 0-72, with higher scores indicating better cognitive function.

SECONDARY OUTCOMES:
Change in appendicular lean mass index | Baseline (M0), 6-month follow-up (M6), 12-month follow-up (M12)
  Change in appendicular lean mass index (ALMI) as measured by dual-energy X-ray absorptiometry (DXA) with higher scores indicating more lean mass. Appendicular lean mass, as measured by DXA, will be divided by height to determine ALMI. ALMI score is a continuous variable with no minimum or maximum value.
Change in physical function | Baseline (M0), 6-month follow-up (M6), 12-month follow-up (M12)
  The Short Physical Performance Battery (SPPB) will be used to assess physical function. Higher scores on the SPPB are indicative of better physical function. The SPPB has a minimum score of 0 and a maximum score of 12.
Change in functional capacity | Baseline (M0), 6-month follow-up (M6), 12-month follow-up (M12)
  The Six Minute Walk Test (6MWT) will be used to measure functional capacity. The 6MWT is scored as distance walked in the 6 minutes with greater distance indicating greater functional capacity.
Change in upper body strength | Baseline (M0), 6-month follow-up (M6), 12-month follow-up (M12)
  Change in grip strength as measured by hand grip dynamometry with higher scores indicating greater upper body strength. Hand grip strength is a continuous variable with no minimum or maximum value.
Change in lower body strength | Baseline (M0), 6-month follow-up (M6), 12-month follow-up (M12)
  Change in quadriceps strength as measured by hand-held quadriceps dynamometry with higher scores indicating greater lower body strength. Quadriceps strength is a continuous variable with no minimum or maximum value.
Change in physical activity | Baseline (M0), 6-month follow-up (M6), 12-month follow-up (M12)
  Change in daily minutes of moderate to vigorous physical activity (MVPA) will be measured via accelerometry with more minutes of daily MVPA indicating more physical activity.
Change in cancer-related fatigue | Baseline (M0), 6-month follow-up (M6), 12-month follow-up (M12)
  The Functional Assessment in Chronic Illness Therapy (FACIT) - Fatigue Scale will be used to measure cancer-related fatigue. Scores range from 0-52, with higher scores indicating less cancer-related fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Diane Ehlers, PhD, Study Director — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will not include identifying information; however, there is still a possibility of deductive disclosure of identity. Therefore, data will not be a shared via an NIH or approved public repository. We will share de-identified as required for publication in scientific journals and with outside collaborators and scientists upon request.
Supporting Information: Study Protocol
Time Frame: Data will be shared via scientific journals at the time of publication and with outside collaborators before publication.
Access Criteria: We will make data available to researchers who agree to use the data only for research purposes, protect the data using secure computer technologies, and destroy the data after relevant analyses are completed and manuscripts are published.